CLINICAL TRIAL: NCT03086369
Title: A Phase 1b (Open-Label) / Phase 2 (Randomized, Double-Blinded) Study Evaluating Nab-Paclitaxel and Gemcitabine With or Without Olaratumab in the Treatment of First-Line Metastatic Pancreatic Cancer
Brief Title: A Study of Nab-Paclitaxel and Gemcitabine With or Without Olaratumab (LY3012207) in Participants With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15844; I5B-MC-JGDP (Other: Eli Lilly and Company); 2016-001099-31 (EudraCT Number)
Record Dates: First submitted 2017-03-13; First posted 2017-03-22 (Actual); Results first posted 2022-01-11 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — olaratumab; 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase1b: Olaratumab 15 mg/kg + Nab-paclitaxel + Gemcitabine (Experimental): Participants received intravenous (IV) infusions of olaratumab 15 milligrams per kilogram (mg/kg), nab-paclitaxel 125 milligrams per meter square (mg/m^2) and gemcitabine 1000 mg/m^2 on days 1, 8, 15 of a 28-day cycle until disease progression or a criterion for discontinuation were met.
  Interventions: Drug: Olaratumab; Drug: Nab-paclitaxel; Drug: Gemcitabine
- Phase1b: Olaratumab 20 mg/kg + Nab-paclitaxel + Gemcitabine (Experimental): Participants received intravenous infusions of olaratumab 20 mg/kg, nab-paclitaxel 125 mg/m^2 and gemcitabine 1000 mg/m^2 on days 1, 8, 15 of a 28-day cycle until disease progression or a criterion for discontinuation were met.
  Interventions: Drug: Olaratumab; Drug: Nab-paclitaxel; Drug: Gemcitabine
- Phase1b (cohort expansion): Olaratumab 20 mg/kg + Nab-paclitaxel + Gemcitabine (Experimental): Following a protocol amendment, "cohort expansion" arm was added in phase 1b with new participants enrolled to confirm the safety of the olaratumab 20 mg/kg dose prior to opening the Phase 2. Participants received intravenous infusions of olaratumab 20 mg/kg, nab-paclitaxel 125 mg/m^2 and gemcitabine 1000 mg/m^2 on days 1, 8, 15 of a 28-day cycle until disease progression or a criterion for discontinuation were met.
  Interventions: Drug: Olaratumab; Drug: Nab-paclitaxel; Drug: Gemcitabine
- Phase 2: Olaratumab + Nab-paclitaxel + Gemcitabine (Experimental): Participants received intravenous infusions of olaratumab 20 mg/kg loading dose on days 1, 8, 15 of cycle 1 followed by 15 mg/kg on days 1, 8, 15 of all subsequent cycles, in combination with nab-paclitaxel 125 mg/m^2 and gemcitabine 1000 mg/m^2 on days 1, 8, 15 of a 28-day cycle until disease progression or a criterion for discontinuation were met.
  Interventions: Drug: Olaratumab; Drug: Nab-paclitaxel; Drug: Gemcitabine
- Phase 2: Placebo + Nab-paclitaxel + Gemcitabine (Placebo Comparator): Participants received intravenous infusions of placebo, nab-paclitaxel 125 mg/m^2 and gemcitabine 1000 mg/m^2 on days 1, 8, 15 of a 28-day cycle until disease progression or a criterion for discontinuation were met.
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine; Drug: Placebo

INTERVENTIONS:
Drug: Olaratumab — Administered IV
  Other Names: LY3012207
  Arms: Phase 2: Olaratumab + Nab-paclitaxel + Gemcitabine; Phase1b (cohort expansion): Olaratumab 20 mg/kg + Nab-paclitaxel + Gemcitabine; Phase1b: Olaratumab 15 mg/kg + Nab-paclitaxel + Gemcitabine; Phase1b: Olaratumab 20 mg/kg + Nab-paclitaxel + Gemcitabine
Drug: Nab-paclitaxel — Administered IV
Drug: Gemcitabine — Administered IV
Drug: Placebo — Administered IV
  Arms: Phase 2: Placebo + Nab-paclitaxel + Gemcitabine

SUMMARY:
The purpose of this study is to determine the safety and efficacy of nab-paclitaxel and gemcitabine with or without olaratumab in the treatment of first-line metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of adenocarcinoma of the exocrine pancreas that is metastatic (Stage IV) and not amenable to resection with curative intent.
* If present, clinically significant or symptomatic amounts of ascites should be drained prior to Day 1.
* Have had no prior systemic treatment for metastatic disease. Prior adjuvant or neo-adjuvant chemotherapy or radiochemotherapy (other than nab-paclitaxel) is allowed if completed ≥3 months prior to enrollment and no lingering toxicities are present.
* Prior radiation therapy for treatment of cancer is allowed to <25% of the bone marrow.
* Phase 2: archival tumor tissue or be willing to provide a pre-treatment biopsy.
* Measurable or nonmeasurable but evaluable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST 1.1).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Discontinued all previous treatments for cancer ≥4 weeks prior.
* Adequate organ function.
* Life expectancy of at least 3 months.

Exclusion Criteria:

* Serious concomitant systemic disorder.
* Have received first line treatment for metastatic pancreatic cancer.
* Received prior treatment with nab-paclitaxel.
* Have known central nervous system malignancy or metastasis.
* Current hematologic malignancies.
* Participated within the last 30 days in a clinical trial involving an investigational product.
* Women with a positive pregnancy test or lactating.
* Have endocrine pancreatic tumors or ampullary cancer.
* Currently enrolled in another clinical trial.
* Have a known additional malignancy that is progressing or required active treatment within the past 1 year.
* Known allergy to nab-paclitaxel or gemcitabine or any ingredient of study drug formulations.
* Are taking certain anti-coagulant medications such as warfarin and are unable to be switched to other similar medicines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (34):
- United States (32):
  - TGen Clinical Research Services at Scottsdale Healthcare, Scottsdale, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - St Jude Medical Center, Fullerton, California
  - TRIO - Translational Research in Oncology-US, Inc., Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Cancer Center of Santa Barbara with Sansum Clinic, Santa Barbara, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists and Research Institute, St. Petersburg, Florida
  - H Lee Moffitt Cancer Center, Tampa, Florida
  - Fort Wayne Oncology & Hematology, Fort Wayne, Indiana
  - Cancer Center of Kansas, Wichita, Kansas
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Monter Cancer Center, Lake Success, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Sanford Research/USD, Sioux Falls, South Dakota
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Sarah Cannon Research Institute SCRI, Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Univ of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah
  - University of Wisconsin-Madison Hospital and Health Clinic, Madison, Wisconsin
- Charité Campus Virchow-Klinikum, Berlin, Germany
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Nab-Paclitaxel and Gemcitabine With or Without Olaratumab (LY3012207) in Participants With Metastatic Pancreatic Cancer — https://trials.lillytrialguide.com/en-US/trial/13wSI7GbbMae4kSSGsoWOw

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers included participants who died from any cause.
Groups:
- Phase1b: Olaratumab 15 mg/kg + Nab-paclitaxel + Gemcitabine: Participants received intravenous infusions of olaratumab 15 milligrams per kilogram (mg/kg), nab-paclitaxel 125 milligrams per meter square (mg/m^2) and gemcitabine 1000 mg/m^2 on days 1, 8, 15 of a 28-day cycle until disease progression or a criterion for discontinuation were met.
Period: Overall Study
Arm/Group | Phase1b: Olaratumab 15 mg/kg + Nab-paclitaxel + Gemcitabine | Phase1b: Olaratumab 20 mg/kg + Nab-paclitaxel + Gemcitabine | Phase1b (Cohort Expansion): Olaratumab 20 mg/kg + Nab-paclitaxel + Gemcitabine | Phase 2: Olaratumab + Nab-paclitaxel + Gemcitabine | Phase 2: Placebo + Nab-paclitaxel + Gemcitabine
Started | 3 | 7 | 12 | 82 | 80
Received at Least 1 Dose of Study Drug | 3 | 7 | 12 | 81 | 78
Completed | 2 | 7 | 12 | 73 | 73
Not Completed | 1 | 0 | 0 | 9 | 7
Not completed — Lost to Follow-up | 1 | 0 | 0 | 2 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 5 | 3
Not completed — Progressive Disease | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All participants in phase 1b/2.
Groups:
- Phase1b: Olaratumab 15 mg/kg + Nab-paclitaxel + Gemcitabine: Participants received intravenous infusions of olaratumab 15 mg/kg, nab-paclitaxel 125 mg/m^2 and gemcitabine 1000 mg/m^2 on days 1, 8, 15 of a 28-day cycle until disease progression or a criterion for discontinuation were met.
- Total: Total of all reporting groups
Arm/Group | Phase1b: Olaratumab 15 mg/kg + Nab-paclitaxel + Gemcitabine | Phase1b: Olaratumab 20 mg/kg + Nab-paclitaxel + Gemcitabine | Phase1b (Cohort Expansion): Olaratumab 20 mg/kg + Nab-paclitaxel + Gemcitabine | Phase 2: Olaratumab + Nab-paclitaxel + Gemcitabine | Phase 2: Placebo + Nab-paclitaxel + Gemcitabine | Total
Number analyzed (Participants) | 3 | 7 | 12 | 82 | 80 | 184
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 3 | 4 | 32 | 37 | 76
  >=65 years | 3 | 4 | 8 | 50 | 43 | 108
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 29 | 35 | 72
  Male | 1 | 4 | 9 | 53 | 45 | 112
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 7 | 8 | 16
  Not Hispanic or Latino | 3 | 7 | 11 | 74 | 70 | 165
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 4 | 3 | 7
  White | 3 | 7 | 12 | 72 | 73 | 167
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 5 | 7 | 76 | 73 | 162
  Germany | 1 | 1 | 5 | 3 | 3 | 13
  Spain | 1 | 1 | 0 | 3 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: A DLT is defined as an adverse event that is likely related to the study medication or combination, and fulfils any one of the following criteria, graded according to the NCI-CTCAE version 4.03:
  1. Any febrile neutropenia
  2. Grade 4 thrombocytopenia, or Grade 3 thrombocytopenia complicated by clinically significant hemorrhage
  3. Grade 4 neutropenia lasting 7 days or longer
  4. Nonhematologic Grade ≥3 toxicity, except for toxicities such as nausea, vomiting, transient electrolyte abnormalities, diarrhea which can be controlled with optimal medical management within 48 hours; non-clinically significant, treatable, or reversible laboratory abnormalities including liver function tests, uric acid, electrolytes, etc.
  5. Any other significant toxicity deemed to be dose-limiting (e.g., any toxicity that is possibly related to the study medication that requires the withdrawal of the participant from the study during Cycle 1).
Time Frame: Cycle 1 (Up to 28 days)
Population: All participants in phase 1b who received at least one dose of Olaratumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase1b: Olaratumab 15 mg/kg + Nab-paclitaxel + Gemcitabine | Phase1b: Olaratumab 20 mg/kg + Nab-paclitaxel + Gemcitabine | Phase1b (Cohort Expansion): Olaratumab 20 mg/kg + Nab-paclitaxel + Gemcitabine
Number analyzed (Participants) | 3 | 7 | 12
Participants | 0 | 0 | 0

2. Primary Outcome: Phase 2: Overall Survival (OS)
Description: OS is defined as the time from the date of randomization to the date of death from any cause. If the participant is alive or lost to follow-up at the time of data analysis, OS data will be censored on the last date the participant is known to be alive. For any participant who has withdrawn consent for further follow-up of survival data, OS will be censored at the last date for which the participant consented to be followed for the study.
Time Frame: Baseline to Date of Death from Any Cause (Up To 29 Months)
Population: All randomized participants in phase 2 (including the censored participants). Number of participants censored in Olaratumab+Nab-paclitaxel+Gemcitabine=26, Placebo+Nab-paclitaxel+Gemcitabine=21.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: Olaratumab + Nab-paclitaxel + Gemcitabine | Phase 2: Placebo + Nab-paclitaxel + Gemcitabine
Number analyzed (Participants) | 82 | 80
Months | 9.10 [7.49 to 14.09] | 10.81 [8.51 to 14.75]
Statistical Analysis 1: Comparison: Phase 2: Olaratumab + Nab-paclitaxel + Gemcitabine vs Phase 2: Placebo + Nab-paclitaxel + Gemcitabine; Test type: Superiority; p = 0.7902, Log Rank; Stratified by age group (<70 years versus ≥70 years) and prior adjuvant/neo-adjuvant gemcitabine use (yes vs no); Hazard Ratio (HR) = 1.054, 95% CI 2-sided [0.728 to 1.527] — Stratified by age group (<70 years versus ≥70 years) and prior adjuvant/neo-adjuvant gemcitabine use (yes vs no)

3. Secondary Outcome: Phase 1b/2: Pharmacokinetics (PK): Minimum Concentration (Cmin) of Olaratumab
Description: PK: Cmin of olaratumab
Time Frame: Pre-dose, 5 min, 1, 4, 4.5, 24, 96, 168, 336 h post-dose on Cycle 1 Day 1, Cycle 1 Day 15, Cycle 3 Day 1, Cycle 3 Day 15
Population: All participants in phase 1b/2 who received at least one dose of Olaratumab and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (μg/mL)
Arm/Group | Phase1b: Olaratumab 15 mg/kg + Nab-paclitaxel + Gemcitabine | Phase1b: Olaratumab 20 mg/kg + Nab-paclitaxel + Gemcitabine | Phase1b (Cohort Expansion): Olaratumab 20 mg/kg + Nab-paclitaxel + Gemcitabine | Phase 2: Olaratumab + Nab-paclitaxel + Gemcitabine
Number analyzed (Participants) | 3 | 5 | 9 | 66
micrograms per milliliter (μg/mL)
  Cycle 1 (Day 1): number analyzed (Participants) | 3 | 5 | 9 | 61
  Cycle 1 (Day 1) | 128 (36) | 86.3 (90) | 87.8 (91) | 112 (40)
  Cycle 1 (Day 15) | 78.7 (42) | 172 (76) | 101 (36) | 94.7 (62)
  Cycle 3 (Day 1): number analyzed (Participants) | 3 | 1 | 9 | 51
  Cycle 3 (Day 1) | 204 (13) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation couldn't be calculated as there was only one participant. Individual value reported: 184 μg/mL | 173 (33) | 147 (38)
  Cycle 3 (Day 15): number analyzed (Participants) | 3 | 1 | 9 | 44
  Cycle 3 (Day 15) | 159 (17) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation couldn't be calculated as there was only one participant. Individual value reported: 99.7 μg/mL | 101 (37) | 106 (68)

4. Secondary Outcome: Phase 2: Number of Participants With Treatment Emergent Anti-Olaratumab Antibodies
Description: Number of Participants With Treatment Emergent Anti-Olaratumab Antibodies
Time Frame: Baseline through Follow-up (Up To 29 Months)
Population: All randomized participants in phase 2 who received at least one dose of Olaratumab and had evaluable immunogenicity data.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Olaratumab + Nab-paclitaxel + Gemcitabine
Number analyzed (Participants) | 81
Participants | 0

5. Secondary Outcome: Phase 1b: Overall Survival (OS)
Description: as for outcome 2
Time Frame: Baseline to Date of Death from Any Cause (Approximately 9 Months)
Population: Phase 1b: Zero participants analysed as data was not collected. OS was not measured in phase 1b.
Arm/Group | Phase1b: Olaratumab 15 mg/kg + Nab-paclitaxel + Gemcitabine | Phase1b: Olaratumab 20 mg/kg + Nab-paclitaxel + Gemcitabine | Phase1b (Cohort Expansion): Olaratumab 20 mg/kg + Nab-paclitaxel + Gemcitabine
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Phase 2: Progression-Free Survival (PFS)
Description: PFS is defined as the time from randomization to the first date of radiologic disease progression (as defined by Response Evaluation Criteria In Solid Tumors, Version 1.1 [RECIST v.1.1]) or death due to any cause in the absence of progressive disease (PD). PD is defined as at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. Participants who did not progress or are lost to follow-up were censored at the day of their last radiographic tumor assessment, if available, or date of randomization if no post-baseline radiographic assessment is available. If death or PD occurs after 2 or more consecutive missing radiographic visits, censoring will occur at the date of the last radiographic visit prior to the missed visits.
Time Frame: Baseline to Disease Progression or Death (Up To 26 Months)
Population: All randomized participants in phase 2 (including the censored participants). Number of participants censored in Olaratumab+Nab-paclitaxel+Gemcitabine=24, Placebo+Nab-paclitaxel+Gemcitabine=26.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: Olaratumab + Nab-paclitaxel + Gemcitabine | Phase 2: Placebo + Nab-paclitaxel + Gemcitabine
Number analyzed (Participants) | 82 | 80
Months | 5.55 [4.14 to 7.0] | 6.41 [5.42 to 7.98]
Statistical Analysis 1: Comparison: Phase 2: Olaratumab + Nab-paclitaxel + Gemcitabine vs Phase 2: Placebo + Nab-paclitaxel + Gemcitabine; Test type: Superiority; p = 0.3771, Log Rank; Stratified by age group (<70 years versus ≥70 years) and prior adjuvant/neo-adjuvant gemcitabine use (yes vs no); Hazard Ratio (HR) = 1.192, 95% CI 2-sided [0.806 to 1.764] — Stratified by age group (<70 years versus ≥70 years) and prior adjuvant/neo-adjuvant gemcitabine use (yes vs no)

7. Secondary Outcome: Phase 1b/2: Objective Response Rate (ORR): Percentage of Participants Who Achieve Complete Response (CR) or Partial Response (PR)
Description: ORR is the best overall tumor response of CR or PR as classified by the investigator according to the Response Evaluation Criteria In Solid Tumors (RECIST v1.1). CR is a disappearance of all target and non-target lesions and normalization of tumor marker level. PR is an at least 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameter) without progression of non-target lesions or appearance of new lesions.
Time Frame: Baseline through Disease Progression or Death (Up To 26 Months)
Population: All participants in phase 1b/2.
Measure: Number; unit: Percentage of participants
Arm/Group | Phase1b: Olaratumab 15 mg/kg + Nab-paclitaxel + Gemcitabine | Phase1b: Olaratumab 20 mg/kg + Nab-paclitaxel + Gemcitabine | Phase1b (Cohort Expansion): Olaratumab 20 mg/kg + Nab-paclitaxel + Gemcitabine | Phase 2: Olaratumab + Nab-paclitaxel + Gemcitabine | Phase 2: Placebo + Nab-paclitaxel + Gemcitabine
Number analyzed (Participants) | 3 | 7 | 12 | 82 | 80
Percentage of participants | 33.3 | 14.3 | 0 | 30.5 | 33.8

8. Secondary Outcome: Phase 1b/2: Duration of Response (DoR)
Description: DoR is defined as the time from the date measurement criteria for CR or PR (whichever is first recorded) are first met until the first date that disease is recurrent or objective progression is observed, per RECIST 1.1 criteria, or the date of death from any cause in the absence of objectively determined disease progression or recurrence.
Time Frame: From Date of CR or PR to Date of Objective Disease Progression or Death Due to Any Cause (Up To 19 Months)
Population: All participants in phase 1b/2 who had CR or PR responses. For phase 1b cohort expansion arm, there were no participants with CR or PR responses to evaluate DoR, hence, zero participants analysed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase1b: Olaratumab 15 mg/kg + Nab-paclitaxel + Gemcitabine | Phase1b: Olaratumab 20 mg/kg + Nab-paclitaxel + Gemcitabine | Phase1b (Cohort Expansion): Olaratumab 20 mg/kg + Nab-paclitaxel + Gemcitabine | Phase 2: Olaratumab + Nab-paclitaxel + Gemcitabine | Phase 2: Placebo + Nab-paclitaxel + Gemcitabine
Number analyzed (Participants) | 1 | 1 | 0 | 25 | 27
Months | NA [NA to NA] — Median and 95% Confidence Interval couldn't be calculated as there was only one participant. Individual value reported: 6.24 months. | NA [NA to NA] — Median and 95% Confidence Interval couldn't be calculated as there was only one participant. Individual value reported: 3.68 months. |  | 5.55 [2.63 to 9.23] | 5.55 [3.84 to 7.26]

9. Secondary Outcome: Phase 2: Time to First Worsening of the Brief Pain Inventory Short Form Modified (mBPI-sf) "Worst Pain Score"
Description: The mBPI-sf is a 11-item instrument used as a multiple-item measure of cancer pain intensity ranging from 0 (no pain or does not interfere) and ranged through 10 (pain as bad as you can imagine or completely interferes). Time to first worsening of the mBPI-sf "worst pain score" (TWP) was defined as the time from the date of randomization to the first date of either a "worst pain" score increase of greater than or equal to (≥) 2 points from baseline or an analgesic drug class increase of ≥1 level. If the participant has not worsened by either of these criteria, TWP was censored for analysis on the last date the mBPI-sf was administered.
Time Frame: Baseline through Follow-up (Up To 21 Months)
Population: All randomized participants in phase 2 who had baseline and at least one post-baseline assessment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: Olaratumab + Nab-paclitaxel + Gemcitabine | Phase 2: Placebo + Nab-paclitaxel + Gemcitabine
Number analyzed (Participants) | 51 | 47
Months | 14.13 [5.19 to NA] — There were not enough events to estimate the upper confidence limit. | 6.11 [2.04 to 9.95]
Statistical Analysis 1: Comparison: Phase 2: Olaratumab + Nab-paclitaxel + Gemcitabine vs Phase 2: Placebo + Nab-paclitaxel + Gemcitabine; Test type: Superiority; p = 0.017, Log Rank; Stratified by age group (<70 years versus ≥70 years) and prior adjuvant/neo-adjuvant gemcitabine use (yes vs no); Hazard Ratio (HR) = 0.390, 95% CI 2-sided [0.175 to 0.872]

10. Secondary Outcome: Phase 2: Time to First Worsening of Symptom Burden on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) - Symptom Scales.
Description: The EORTC QLQ-C30 is a self-reported general cancer instrument consisting of 30 items covered by 1 of 3 dimensions: global health status/quality of life (2 items), functional scales (15 total items addressing either physical, role, emotional, cognitive, or social functioning), symptom scales (13 total items addressing either fatigue, nausea/vomiting, pain, dyspnoea, insomnia, appetite loss, constipation, diarrhoea, or financial impact). Time to first worsening of Symptom Burden was defined as the time from randomization to the first observation of worsening on symptom scales (i.e.,) increase of at least 10 points from baseline. For symptom scales, a linear transformation was used to obtain total score ranging from 0 to 100, a high score represents a high level of symptomatology or problems.
Time Frame: Baseline through Follow-up (Up To 21 Months)
Population: All randomized participants in phase 2 who had baseline and at least one post-baseline assessment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: Olaratumab + Nab-paclitaxel + Gemcitabine | Phase 2: Placebo + Nab-paclitaxel + Gemcitabine
Number analyzed (Participants) | 68 | 66
Months
  Appetite loss: number analyzed (Participants) | 57 | 60
  Appetite loss | NA [2.79 to NA] — There were not enough events to estimate median, upper confidence limit. | 2.86 [1.94 to NA] — There were not enough events to estimate upper confidence limit.
  Constipation: number analyzed (Participants) | 64 | 59
  Constipation | NA [2.76 to NA] — There were not enough events to estimate median, upper confidence limit. | NA [1.94 to NA] — There were not enough events to estimate median, upper confidence limit.
  Diarrhoea: number analyzed (Participants) | 68 | 62
  Diarrhoea | 2.79 [1.87 to NA] — There were not enough events to estimate upper confidence limit. | 1.97 [1.91 to NA] — There were not enough events to estimate upper confidence limit.
  Dyspnoea: number analyzed (Participants) | 66 | 66
  Dyspnoea | 2.79 [2.10 to NA] — There were not enough events to estimate upper confidence limit. | 3.12 [2.07 to NA] — There were not enough events to estimate upper confidence limit.
  Fatigue: number analyzed (Participants) | 66 | 64
  Fatigue | 1.87 [1.05 to 2.33] | 1.87 [1.12 to 2.07]
  Financial difficulties: number analyzed (Participants) | 65 | 61
  Financial difficulties | NA [2.37 to NA] — There were not enough events to estimate median, upper confidence limit. | NA [2.79 to NA] — There were not enough events to estimate median, upper confidence limit.
  Insomnia: number analyzed (Participants) | 60 | 60
  Insomnia | 3.19 [2.10 to NA] — There were not enough events to estimate upper confidence limit. | NA [2.83 to NA] — There were not enough events to estimate median, upper confidence limit.
  Nausea and vomiting: number analyzed (Participants) | 66 | 66
  Nausea and vomiting | 3.19 [2.10 to NA] — There were not enough events to estimate upper confidence limit. | 2.86 [1.97 to NA] — There were not enough events to estimate upper confidence limit.
  Pain: number analyzed (Participants) | 64 | 58
  Pain | NA [2.76 to NA] — There were not enough events to estimate median, upper confidence limit. | 3.25 [2.04 to NA] — There were not enough events to estimate upper confidence limit.
Statistical Analysis 1: Comparison: Phase 2: Olaratumab + Nab-paclitaxel + Gemcitabine vs Phase 2: Placebo + Nab-paclitaxel + Gemcitabine; Appetite loss; Test type: Superiority; p = 0.288, Log Rank; Stratified by age group (<70 years versus ≥70 years) and prior adjuvant/neo-adjuvant gemcitabine use (yes vs no); Hazard Ratio (HR) = 0.718, 95% CI 2-sided [0.392 to 1.317] — Stratified by age group (<70 years versus ≥70 years) and prior adjuvant/neo-adjuvant gemcitabine use (yes vs no)
Statistical Analysis 2: Comparison: Phase 2: Olaratumab + Nab-paclitaxel + Gemcitabine vs Phase 2: Placebo + Nab-paclitaxel + Gemcitabine; Constipation; Test type: Superiority; p = 0.442, Log Rank; Stratified by age group (<70 years versus ≥70 years) and prior adjuvant/neo-adjuvant gemcitabine use (yes vs no); Hazard Ratio (HR) = 0.788, 95% CI 2-sided [0.423 to 1.468] — Stratified by age group (<70 years versus ≥70 years) and prior adjuvant/neo-adjuvant gemcitabine use (yes vs no)
Statistical Analysis 3: Comparison: Phase 2: Olaratumab + Nab-paclitaxel + Gemcitabine vs Phase 2: Placebo + Nab-paclitaxel + Gemcitabine; Diarrhoea; Test type: Superiority; p = 0.883, Log Rank; Stratified by age group (<70 years versus ≥70 years) and prior adjuvant/neo-adjuvant gemcitabine use (yes vs no); Hazard Ratio (HR) = 1.037, 95% CI 2-sided [0.612 to 1.755] — Stratified by age group (<70 years versus ≥70 years) and prior adjuvant/neo-adjuvant gemcitabine use (yes vs no)
Statistical Analysis 4: Comparison: Phase 2: Olaratumab + Nab-paclitaxel + Gemcitabine vs Phase 2: Placebo + Nab-paclitaxel + Gemcitabine; Dyspnoea; Test type: Superiority; p = 0.803, Log Rank; Stratified by age group (<70 years versus ≥70 years) and prior adjuvant/neo-adjuvant gemcitabine use (yes vs no); Hazard Ratio (HR) = 0.933, 95% CI 2-sided [0.532 to 1.636] — Stratified by age group (<70 years versus ≥70 years) and prior adjuvant/neo-adjuvant gemcitabine use (yes vs no)
Statistical Analysis 5: Comparison: Phase 2: Olaratumab + Nab-paclitaxel + Gemcitabine vs Phase 2: Placebo + Nab-paclitaxel + Gemcitabine; Fatigue; Test type: Superiority; p = 0.805, Log Rank; Stratified by age group (<70 years versus ≥70 years) and prior adjuvant/neo-adjuvant gemcitabine use (yes vs no); Hazard Ratio (HR) = 1.053, 95% CI 2-sided [0.675 to 1.645] — Stratified by age group (<70 years versus ≥70 years) and prior adjuvant/neo-adjuvant gemcitabine use (yes vs no)
Statistical Analysis 6: Comparison: Phase 2: Olaratumab + Nab-paclitaxel + Gemcitabine vs Phase 2: Placebo + Nab-paclitaxel + Gemcitabine; Financial difficulties; Test type: Superiority; p = 0.465, Log Rank; Stratified by age group (<70 years versus ≥70 years) and prior adjuvant/neo-adjuvant gemcitabine use (yes vs no); Hazard Ratio (HR) = 0.784, 95% CI 2-sided [0.420 to 1.464] — Stratified by age group (<70 years versus ≥70 years) and prior adjuvant/neo-adjuvant gemcitabine use (yes vs no)
Statistical Analysis 7: Comparison: Phase 2: Olaratumab + Nab-paclitaxel + Gemcitabine vs Phase 2: Placebo + Nab-paclitaxel + Gemcitabine; Insomnia; Test type: Superiority; p = 0.231, Log Rank; Stratified by age group (<70 years versus ≥70 years) and prior adjuvant/neo-adjuvant gemcitabine use (yes vs no); Hazard Ratio (HR) = 1.457, 95% CI 2-sided [0.787 to 2.698] — Stratified by age group (<70 years versus ≥70 years) and prior adjuvant/neo-adjuvant gemcitabine use (yes vs no)
Statistical Analysis 8: Comparison: Phase 2: Olaratumab + Nab-paclitaxel + Gemcitabine vs Phase 2: Placebo + Nab-paclitaxel + Gemcitabine; Nausea and vomiting; Test type: Superiority; p = 0.748, Log Rank; Stratified by age group (<70 years versus ≥70 years) and prior adjuvant/neo-adjuvant gemcitabine use (yes vs no); Hazard Ratio (HR) = 0.914, 95% CI 2-sided [0.532 to 1.570] — Stratified by age group (<70 years versus ≥70 years) and prior adjuvant/neo-adjuvant gemcitabine use (yes vs no)
Statistical Analysis 9: Comparison: Phase 2: Olaratumab + Nab-paclitaxel + Gemcitabine vs Phase 2: Placebo + Nab-paclitaxel + Gemcitabine; Pain; Test type: Superiority; p = 0.875, Log Rank; Stratified by age group (<70 years versus ≥70 years) and prior adjuvant/neo-adjuvant gemcitabine use (yes vs no); Hazard Ratio (HR) = 0.947, 95% CI 2-sided [0.491 to 1.827] — Stratified by age group (<70 years versus ≥70 years) and prior adjuvant/neo-adjuvant gemcitabine use (yes vs no)

11. Secondary Outcome: Phase 2: Health Status on the EuroQol 5-Dimension 5 Level (EQ-5D-5L)
Description: The EQ-5D-5L is a standardized instrument for use as a measure of self-reported health status. Five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) of health status are each assessed with 5 response options (1=no problem, 2=slight, 3=moderate, 4=severe, and 5=extreme problem) and scored as a composite index which were anchored on a scale of 0 to 1 with a higher score representing better health status. Additionally, current health status was assessed on a visual analogue scale (VAS) ranging from 0 to 100 with a higher score representing better health status.
Time Frame: Cycle 1 Day 1, Cycle 7 Day 1
Population: All randomized participants in phase 2 who completed EQ-5D-5L.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2: Olaratumab + Nab-paclitaxel + Gemcitabine | Phase 2: Placebo + Nab-paclitaxel + Gemcitabine
Number analyzed (Participants) | 70 | 70
score on a scale
  Index Value [Cycle 1 (Day1)]: number analyzed (Participants) | 69 | 70
  Index Value [Cycle 1 (Day1)] | 0.8 (0.2) | 0.8 (0.2)
  Index Value [Cycle 7 (Day1)]: number analyzed (Participants) | 22 | 33
  Index Value [Cycle 7 (Day1)] | 0.8 (0.1) | 0.8 (0.2)
  VAS Score [Cycle 1 (Day1)] | 70.1 (21.7) | 69.7 (20.4)
  VAS Score [Cycle 7 (Day1)]: number analyzed (Participants) | 23 | 33
  VAS Score [Cycle 7 (Day1)] | 71.7 (20.2) | 73.2 (22.5)

ADVERSE EVENTS:
Time Frame: Baseline to Follow-up (Up To 29 Months)
Description: All participants in phase 1b/2 who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | Phase1b: Olaratumab 15 mg/kg + Nab-paclitaxel + Gemcitabine | Phase1b: Olaratumab 20 mg/kg + Nab-paclitaxel + Gemcitabine | Phase1b (Cohort Expansion): Olaratumab 20 mg/kg + Nab-paclitaxel + Gemcitabine | Phase 2: Olaratumab + Nab-paclitaxel + Gemcitabine | Phase 2: Placebo + Nab-paclitaxel + Gemcitabine
All-Cause Mortality (participants affected / at risk) | 2/3 | 7/7 | 12/12 | 60/81 | 63/78
Serious Adverse Events (participants affected / at risk) | 3/3 | 3/7 | 8/12 | 50/81 | 41/78
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 12/12 | 79/81 | 78/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase1b: Olaratumab 15 mg/kg + Nab-paclitaxel + Gemcitabine (N=3) | Phase1b: Olaratumab 20 mg/kg + Nab-paclitaxel + Gemcitabine (N=7) | Phase1b (Cohort Expansion): Olaratumab 20 mg/kg + Nab-paclitaxel + Gemcitabine (N=12) | Phase 2: Olaratumab + Nab-paclitaxel + Gemcitabine (N=81) | Phase 2: Placebo + Nab-paclitaxel + Gemcitabine (N=78)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Amaurosis fugax (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (2) | 5 (5) | 4 (4)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colonic abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device related bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 8 (9)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 2 (2)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drain site complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin b12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Embolic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal cavity drainage (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Phase1b: Olaratumab 15 mg/kg + Nab-paclitaxel + Gemcitabine (N=3) | Phase1b: Olaratumab 20 mg/kg + Nab-paclitaxel + Gemcitabine (N=7) | Phase1b (Cohort Expansion): Olaratumab 20 mg/kg + Nab-paclitaxel + Gemcitabine (N=12) | Phase 2: Olaratumab + Nab-paclitaxel + Gemcitabine (N=81) | Phase 2: Placebo + Nab-paclitaxel + Gemcitabine (N=78)
Anaemia (Blood and lymphatic system disorders) | 2 (8) | 2 (7) | 5 (9) | 46 (186) | 45 (165)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (13) | 1 (2) | 3 (6) | 20 (53) | 16 (70)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (5) | 1 (3) | 5 (6) | 7 (19) | 12 (93)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (3)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 4 (5)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 6 (12) | 15 (21) | 16 (22)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 5 (7)
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (4) | 4 (5) | 22 (26) | 30 (31)
Diarrhoea (Gastrointestinal disorders) | 2 (4) | 1 (1) | 7 (9) | 40 (72) | 30 (58)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (5)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (6)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 6 (15) | 33 (46) | 39 (62)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 9 (11) | 9 (11)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (4) | 19 (26) | 19 (23)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (2) | 11 (12) | 10 (18)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 8 (10) | 12 (17)
Fatigue (General disorders) | 2 (10) | 3 (4) | 9 (19) | 53 (74) | 44 (84)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 5 (14)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (4)
Oedema peripheral (General disorders) | 2 (4) | 0 (0) | 5 (8) | 25 (43) | 28 (44)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Pyrexia (General disorders) | 0 (0) | 1 (2) | 1 (1) | 20 (30) | 21 (28)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergy to arthropod bite (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 4 (4) | 3 (8)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 5 (5)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Skin infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 3 (7) | 2 (5)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 8 (16)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) | 1 (1) | 3 (4) | 6 (6)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 5 (6)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 13 (28) | 14 (26)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 15 (38) | 13 (20)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 8 (23) | 9 (20)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 8 (12) | 9 (11)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 5 (10)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 3 (13) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 12 (88) | 7 (34)
Neutrophil count decreased (Investigations) | 2 (4) | 3 (15) | 4 (11) | 31 (184) | 25 (128)
Platelet count decreased (Investigations) | 1 (3) | 2 (3) | 3 (9) | 29 (134) | 31 (106)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 2 (2) | 23 (36) | 9 (14)
White blood cell count decreased (Investigations) | 0 (0) | 2 (2) | 3 (5) | 23 (127) | 16 (92)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 22 (26) | 24 (37)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 14 (20) | 15 (30)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 4 (10)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 13 (60) | 4 (7)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 10 (13) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (4) | 19 (40) | 17 (31)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 16 (27) | 12 (20)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 3 (4) | 15 (41) | 6 (11)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2) | 0 (0) | 2 (3) | 7 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 6 (6) | 11 (13)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 4 (5)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 11 (14) | 4 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 8 (8) | 8 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 9 (10) | 6 (11)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 20 (26) | 21 (30)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 8 (11) | 13 (15)
Formication (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 6 (9) | 10 (11)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 4 (4)
Neuropathy peripheral (Nervous system disorders) | 1 (3) | 0 (0) | 3 (9) | 18 (36) | 12 (23)
Neurotoxicity (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 3 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (4) | 0 (0) | 15 (29) | 17 (30)
Polyneuropathy (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 8 (11)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 7 (9) | 5 (7)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (3) | 10 (11) | 11 (13)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1/2 (1) | 0/3 (0) | 0/3 (0) | 0/29 (0) | 0/35 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 13 (14) | 10 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 14 (17) | 13 (25)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0) | 4 (4) | 8 (10)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 4 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 6 (7) | 28 (34) | 16 (21)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (4) | 6 (9) | 13 (22)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (6) | 7 (8)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (4) | 0 (0)
Central venous catheterisation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental implantation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic pseudocyst drainage (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 4 (4)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 7 (14) | 4 (6)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 2 (2) | 14 (18) | 6 (7)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/69/NCT03086369/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-03): https://cdn.clinicaltrials.gov/large-docs/69/NCT03086369/SAP_001.pdf